CLINICAL TRIAL: NCT03285802
Title: CRAD001X2401: Treatment Plan for an Individual Patient With Recurrent Uterine Papillary Serous Carcinoma (UPSC) With PIK3CA Gene Mutation
Brief Title: Treatment Plan for an Individual Patient With Recurrent Uterine Papillary Serous Carcinoma (UPSC) With PIK3CA Gene Mutation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Greater Baltimore Medical Center (Other)
Responsible Party: Principal Investigator, Melissa Loomis, CCRP, Gynecologic Oncologist, Greater Baltimore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001X2401
Record Dates: First submitted 2017-09-07; First posted 2017-09-18 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms | interventions — Letrozole; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Letrozole and Everolimus (Experimental): Letrozole 2.5mg daily q 30 days Everolimus 10mg daily q 28 days
  Interventions: Drug: Letrozole; Drug: Everolimus

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5mg will be taken daily q 30 days
  Other Names: Femara
Drug: Everolimus — Everolimus 10mg daily q 28 days
  Other Names: Afinitor

SUMMARY:
This is an open-label treatment program following basic prescribing information for patients with recurrent UPSC (Uterine Papillary Serous Carcinoma) to provide access to everolimus and limited treatment alternatives.

DETAILED DESCRIPTION:
The objective is to provide access to everolimus for patients with Recurrent UPSC and limited treatment alternatives.

Letrozole 2.5mg daily q 30 days Everolimus 10mg daily q 28 days

ELIGIBILITY:
Inclusion Criteria:

1. Patient has adequate bone marrow and coagulation function as shown by: absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelets ≥ 100 × 109/L; hemoglobin (Hgb) ≥ 9.0 g/dL.
2. Patient has adequate liver function as shown by:

   1. total serum bilirubin ≤2.0 mg/dL,
   2. ALT and AST ≤2.5x ULN (≤5x ULN in patients with liver metastases),
   3. INR ≤2;.
3. Patient has adequate renal function as shown by serum creatinine ≤ 1.5 × ULN.
4. Patient has fasting serum cholesterol ≤ 300mg/dl or 7.75mmol/L AND fasting triglycerides ≤ 2.5 × ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
5. Patient will give a written informed consent obtained according to local guidelines.
6. Sexually active males must use a condom during intercourse while taking everolimus for treatment, for 8 weeks after stopping treatment, or their female partners should use highly effective contraception during this specified time period.
7. Women of childbearing potential must have had a negative serum pregnancy test 14 days prior to the start of everolimus treatment plus a negative local urine pregnancy test prior to treatment and must be willing to use highly effective methods of contraception during the study and for 8 weeks after study drug administration.

Exclusion Criteria:

1. Patient has had prior therapy with mTOR inhibitors (e.g. sirolimus, temsirolimus, deforolimus).
2. Patient has a known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus).
3. Patient has uncontrolled diabetes mellitus as defined by fasting serum glucose > 1.5 × ULN despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout participation in the program and adjusted as necessary.
4. Patient has any severe and/or uncontrolled medical conditions such as:

   1. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to randomization, serious uncontrolled cardiac arrhythmia,
   2. active or uncontrolled severe infection,
   3. liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA),
   4. known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air),
   5. active, bleeding diathesis.
5. Chronic treatment with corticosteroids or other immunosuppressive agents.
6. Patient has a known history of HIV seropositivity.
7. Patient is a woman of child-bearing potential, unless she is using highly effective contraception methods.

   * Women of child-bearing potential (WOCBP) is defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partner has been sterilized by vasectomy or other means.
   * Highly effective contraception, defined as one that results in an annual pregnancy rate <1% when used correctly, comprises one of the following methods:
   * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception)
   * Male/female sterilization
   * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
8. Patient is unwilling to or unable to comply with the treatment plan.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 1 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Single Arm Trial With Combination of Everolimus and Letrozole in Treatment With Recurrent Uterine Papillary Serous Carcinoma (UPSC) With PIK3CA Gene Mutation; Tumor Response to treatment with Everolimus and Letrozole using RECIST Criteria | Baseline, Then every 12 weeks while on Everolimus and Letrozole up to 36 months;
  Tumor Response to treatment with Everolimus and Letrozole using RECIST Criteria

SECONDARY OUTCOMES:
Single Arm Trial With Combination of Everolimus and Letrozole in Treatment With Recurrent Uterine Papillary Serous Carcinoma (UPSC) With PIK3CA Gene Mutation; Overall survival of patients treated with the combination of letrozole and everolimus | From randomization until date of death, assessed up to 36 months
  Overall survival of patients treated with the combination of letrozole and everolimus

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Baltimore Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided